CLINICAL TRIAL: NCT05514613
Title: Comparative Effectiveness of Reel-time Ultrasound-guided Tracheostomy and Anatomic Landmark Percutaneous Dilatational Tracheostomy: a Retrospective Cohort Study
Brief Title: Effectiveness of Reel-time Ultrasound-guided Tracheostomy and Landmark Percutaneous Dilatational Tracheostomy
Status: Completed | Type: Observational
Sponsor: HULYA TOPCU (Other)
Collaborators: Serhat Ozciftci (Unknown)
Responsible Party: Sponsor-Investigator, HULYA TOPCU, assistant professor doctor Hulya TOPCU, Erol Olcok Corum Training and Research Hospital
Organization: Erol Olcok Corum Training and Research Hospital (Other)
Other Study IDs: CorumTRH
Record Dates: First submitted 2022-08-09; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Tracheostomy Complication
Keywords: ultrasound guided tracheostomy; anatomic landmark tracheostomy; tracheostomy; complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group G: Group G is a tracheostomy group opened using the anatomical sign technique (Griggs technique).
  Interventions: Other: retrospektif study; The effect of tracheostomy tecnique method on complications
- Group U: Group U; Ultrasound-guided is used during tracheostomy technique.
  Interventions: Other: retrospektif study; The effect of tracheostomy tecnique method on complications

INTERVENTIONS:
Other: retrospektif study; The effect of tracheostomy tecnique method on complications — retrospektif study; The effect of tracheostomy tecnique method on complications complications and correlation of complications with techniques

SUMMARY:
This study aims to assess the impact of real-time ultrasound (US) use on complication rates and procedural success in percutaneous dilational tracheostomy (PDT) opened with forceps dilatation technique using anatomical landmarks.

DETAILED DESCRIPTION:
This study, patients who were admitted to the intensive care unit of hospital and who had a tracheostomy were examined. This is a retrospective study conducted to evaluate the method used during tracheostomy and themcomplications that occurred during and after tracheostomy opening.

2852 intensive care patients hospitalized in hospital intensive care unit after obtaining ethical permission were investigated retrospectively by scanning their files and digital data, and their complications during and after tracheostomy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in the intensive care unit and tracheostomy was opened and over 18 years.

Exclusion Criteria:

* surgical opened tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who were hospitalized in the intensive care unit and underwent tracheostomy
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Ultrasound-guided Tracheostomy and Landmark Percutaneous Dilatational Tracheostomy | 01.04.2017-11.03.2019
  the relationship of complications with the tracheostomy technique

CONTACTS AND LOCATIONS:
Locations (1):
- Çorum training and research state hospital, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No